CLINICAL TRIAL: NCT01439087
Title: Pilot Study to Evaluate Optical Frequency Domain Imaging as a Tool for Assessing Colonic Polyps
Brief Title: Optical Frequency Domain Imaging for Assessing Colonic Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2009-P000946
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Colonic Polyps
Keywords: Colonic Polyps; OCT; Imaging; Colon; Polyp
MeSH Terms: conditions — Colonic Polyps; Polyps | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OFDI imaging (Experimental): OFDI imaging
  Interventions: Device: MGH Optical Frequency Domain Imaging (OFDI) System

INTERVENTIONS:
Device: MGH Optical Frequency Domain Imaging (OFDI) System — Imaging of Colonic Polyps with OFDI system

SUMMARY:
The goal of this research is to conduct a pilot clinical study to image colonic polyps with the intent to evaluate the potential use of Optical Frequency Domain Imaging (OFDI) to identify the extent of invasion (if present), differentiate between hyperplastic polyps and adenomas, and identify serrated polyps.

DETAILED DESCRIPTION:
The colon OFDI catheter will be used in conjunction with a sigmoidoscope. If a sigmoid polyp is identified, the colonoscope will be removed and a sigmoidoscope inserted. The colon OFDI catheter will be advanced through the sigmoidoscope accessory port and positioned adjacent to the colon wall. Imaging will be performed with the OFDI system across the polyp's surface and the base/stalk if pedunculated. The investigators anticipate that on average the investigators will utilize 4 helical scans per polyp. Each of the scans will take less than 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a screening colonoscopy
* Patients must be over the age of 18
* Patient must be able to give informed consent

Exclusion Criteria:

* Patients with hemostasis disorders
* Patients taking any anti-coagulants such as Coumadin or Plavix,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OFDI Imaging
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OFDI Imaging
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Sensitivity of OFDI Imaging in the Colon
Description: OFDI Images are analyzed and compared to standard of care biopsies in order to differentiate hyperplastic polyps from adenomas or to identify serrated polyps. A total of 15 subjects were consented, but upon inspection of the colon only 2 participants met the eligibility criteria and participated.
Time Frame: During the OFDI imaging session which should take an average of 5 mintues
Measure: Count of Participants; unit: Participants
Groups:
- Feasibility & Sensitivity of OFDI Imaging in the Colon: Feasibility is measured by the number of enrolled subjects that met imaging eligibility criteria and were successfully imaged with the OFDI device.
  Sensitivity is measured by the number of enrolled subjects that met eligibility criteria, and had a polyp(s) successfully imaged and identified by the OFDI device.
Arm/Group | Feasibility & Sensitivity of OFDI Imaging in the Colon
Number analyzed (Participants) | 2
Participants
  Feasibility | 2
  Sensitivity | 1

ADVERSE EVENTS:
Arm/Group | OFDI Imaging
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No